CLINICAL TRIAL: NCT02529293
Title: A Pilot Clinical Trial Investigating the Intra-subject Variability of Pharmacokinetics and Glucodynamics of BioChaperone Insulin Lispro U-100 Product (2 Single Doses of 0.2 U/kg) and U-200 Product (2 Single Doses of 0.2 U/kg) in Healthy Male and Female
Brief Title: A Clinical Trial Investigating the Intra-subject Variability of Pharmacokinetics and Glucodynamics of BioChaperone Insulin Lispro U-100 Product and U-200 Product in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT012
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone Lispro U-100 (Active Comparator): injection of 2 doses of 0.2 U/kg on separate visits
  Interventions: Drug: BioChaperone Lispro U-100
- BioChaperone Lispro U-200 (Experimental): injection of 2 doses of 0.2 U/kg on separate visits
  Interventions: Drug: BioChaperone Lispro U-200

INTERVENTIONS:
Drug: BioChaperone Lispro U-100 — Injection of BioChaperone Lispro U-100
  Arms: BioChaperone Lispro U-100
Drug: BioChaperone Lispro U-200 — Injection of BioChaperone Lispro U-200
  Arms: BioChaperone Lispro U-200

SUMMARY:
This is a double-blinded, randomised, single-centre phase I pilot trial for exploring the feasibility of a pivotal clinical trial establishing bioequivalence between BioChaperone insulin lispro U-200 and BioChaperone insulin lispro U-100 in healthy subjects.

Each subject will be randomly allocated to a sequence of four treatments, i.e. two single doses of BioChaperone insulin lispro U-200 of 0.2 U·kg BW-1 and two single doses of BioChaperone insulin lispro U-100 of 0.2 U·kg BW-1 on four separate dosing visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
* Age ≥ 18 and ≤ 64 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 28.0 kg∙m-2, both inclusive.
* Fasting Plasma Glucose (FPG) ≤ 5.6 mmol/L (100 mg/dL).
* Signed and dated informed consent obtained before any trial-related activities, i.e. any procedures that would not have been performed during normal management of the subject).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Receipt of any investigational medicinal product within 3 months before randomisation in this trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
AUCLisp (0-inf) | 8 hours
  Area under the insulin lispro serum concentration - time curve from t=0 to infinity
Cmax Lisp | 8 hours
  Maximum observed insulin lispro serum concentration

SECONDARY OUTCOMES:
tmax Lisp | 8 hours
  Time to maximum observed serum insulin lispro concentration
AUCGIR(0-8h) | 8 hours
  Area under the glucose infusion rate-time curve from t=0 to 8 hours
GIRmax | 8 hours
  Maximum glucose infusion rate
tGIRmax | 8 hours
  Time to maximum glucose infusion rate
Number of Adverse events | Up to 9 weeks
  Number of adverse events
Local tolerability | Up to 9 weeks
  Record of injection site reaction

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut Für Stoffwechselfforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany